CLINICAL TRIAL: NCT05347888
Title: How Well do we Feed the Critically Ill Patients: a Multicentric, Prospective Observational Study
Brief Title: How Well do we Feed the Critically Ill Patients
Acronym: WE-FEED
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Collaborators: Banaras Hindu University (Other); All India Institute of Medical Sciences (Other); All India Institute of Medical Sciences, Raipur (Other Government); Artemis Hospital, Gurugram, India (Unknown); Atal Bihari Vajpayee Institute of Medical Sciences and Dr RML Hospital, Delhi, India (Unknown); Dr Bhubaneswar Borooah Cancer Hospital, Guwahati, India (Unknown); Father Muller Medical College (Other); Fortis Hospital, India (Other); Govind Ballabh Pant Institute of Postgraduate Medical Education and Research (Other Government); Mata Chanan Devi Hospital, Delhi, India (Unknown); North Eastern Indira Gandhi Regional Institute of Health ans Medical Sciences (Other Government); Rajiv Gandhi Cancer Institute & Research Center, India (Other); Mediclinic Parkview Hospital, Dubai, United Arab Emirates (Unknown); Amina Hospital, Ajman, United Arab Emirates (Unknown); Sri Guru Ram Institute of Medical & Health Science Shri Mahant Indiresh Hospital, Dehradun, India (Unknown)
Responsible Party: Principal Investigator, Prashant Nasa, HOD, Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: NMCSHFeeding
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Enteral and Supplement Feeds Adverse Reaction; Nutrition Deficiency Due to Insufficient Food; Critically Ill; Parenteral Nutrition Associated Liver Disease; Feeding Patterns
MeSH Terms: conditions — Critical Illness; Feeding Behavior | interventions — Nutrition Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nutritional therapy — Either enteral or parenteral nutrition is used for the patient admitted in the ICU

SUMMARY:
The present prospective observational multicentric study will assess the nutritional status of critically ill patients, cumulative calorie and protein balance and the effect of calorie and protein balance on clinical outcomes.

DETAILED DESCRIPTION:
Nutritional therapy is a very important aspect of the management of critically ill patients. These patients need intensive monitoring, various organ supports in the form of vasopressors and inotropes, mechanical ventilation, dialysis, extracorporeal organ supports, infection controls, etc. In this very complex, critical and demanding scenario, nutritional therapy often gets a back seat in the initial period at least till the time patient is stabilised. But this nutritional deprivation has much more deleterious effects in sepsis and systemic inflammatory response syndromes induced catabolic state than that of fasting in healthy persons. Various studies showed that inadequate feeding has been associated with an increased hospital length of stay, incidence of complications, infections, incidence of organ failure, and risk of mortality. A single centre prospective study that analyzed 768 patients reported that 69% were calorie deficient and 90% were protein deficient. They also observed a positive correlation between calorie deficit and infectious complications, length of Intensive Care Unit (ICU) stay and days of mechanical ventilation.

The main factors may hinder enteral feeding and adequate nutrition delivery. That includes delay in the initiation of Enteral Nutrition (EN) and slow infusion rate; low adherence to EN practice guidelines; frequent disruptions to EN due to diagnostic or therapeutic procedures.

In observational studies, patients in the ICU who were fed early through the enteral route have had a better outcome than those who were not. Similarly, overfeeding has also been associated with various complications, including hyperglycemia, hypertriglyceridemia, hepatic steatosis, azotemia, hypercapnia, and an increased rate of mortality among patients.

Therefore, optimum nutrition is vital to a patient's survival. The present prospective observational multicentric study will assess the nutritional status of critically ill patients, cumulative calorie and protein balance and the effect of calorie and protein balance on clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who receive either enteral or parenteral nutrition will be included in the study.

Exclusion Criteria:

* Age less than 18 years old
* Pregnant women
* Patient is expected to die within 48 hours of ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who are treated in the intensive care unit and receive either enteral or parenteral nutrition will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Calorie and protein balance | From day of randomization till 7 days, or the patient is discharged from ICU, or death of the patient, whichever is earlier.
  Cumulative calorie and protein balance.

SECONDARY OUTCOMES:
Length of ICU stay | From the day of randomization till the patient is shifted out of ICU, or death of the patient, or 28 days of ICU admission, whichever is earlier.
  Correlation between initial nutritional status and calorie and protein deficit with length of ICU stay
Days of Mechanical Ventilation | From day of randomization till the patient is removed from mechanical ventilation, or 28 days of ICU admission, or death of the patient, whichever is earlier
  correlation between initial nutritional status and calorie and protein deficit with days of mechanical ventilation
Mortality | From the day of randomisation to 28 days of ICU admission.
  Correlation between initial nutritional status and calorie and protein deficit with mortality
Time to initiation of enteral or parenteral nutrition | From the day of randomisation till 28 days of ICU admission, or death of the patient, whichever is earlier
  Time from ICU admission to initiation of enteral or parenteral nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh K Das, MD, Principal Investigator — Artemis Hospital, Gurugram, India
Locations (1):
- NMC Specialty Hospital, Al Nahda, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloomer MJ, Clarke AB, Morphet J. Nurses' prioritization of enteral nutrition in intensive care units: a national survey. Nurs Crit Care. 2018 May;23(3):152-158. doi: 10.1111/nicc.12284. Epub 2017 Jan 30. PMID 28133862
- [Background] Ventura AM, Waitzberg DL. Enteral nutrition protocols for critically ill patients: are they necessary? Nutr Clin Pract. 2015 Jun;30(3):351-62. doi: 10.1177/0884533614547765. Epub 2014 Sep 23. PMID 25249598
- [Background] Weijs PJ, Looijaard WG, Beishuizen A, Girbes AR, Oudemans-van Straaten HM. Early high protein intake is associated with low mortality and energy overfeeding with high mortality in non-septic mechanically ventilated critically ill patients. Crit Care. 2014 Dec 14;18(6):701. doi: 10.1186/s13054-014-0701-z. PMID 25499096
- [Result] Faisy C, Lerolle N, Dachraoui F, Savard JF, Abboud I, Tadie JM, Fagon JY. Impact of energy deficit calculated by a predictive method on outcome in medical patients requiring prolonged acute mechanical ventilation. Br J Nutr. 2009 Apr;101(7):1079-87. doi: 10.1017/S0007114508055669. Epub 2008 Sep 9. PMID 18778528
- [Result] Giner M, Laviano A, Meguid MM, Gleason JR. In 1995 a correlation between malnutrition and poor outcome in critically ill patients still exists. Nutrition. 1996 Jan;12(1):23-9. doi: 10.1016/0899-9007(95)00015-1. PMID 8838832
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131